CLINICAL TRIAL: NCT05645432
Title: An Open-Label Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of Brexanolone in the Treatment of Adult Participants With Tinnitus
Brief Title: An Open-Label Study Evaluating Brexanolone in Adults With Tinnitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 547-TRM-201
Record Dates: First submitted 2022-12-01; First posted 2022-12-09 (Actual); Results first posted 2024-12-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2024-11

CONDITIONS: Tinnitus
Keywords: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — brexanolone; Pregnanolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexanolone (Experimental): Participants will receive a 6-hour single continuous intravenous (IV) infusion of brexanolone at 30 micrograms per kilogram per hour (mcg/kg/hour) for 0 to 0.5 hours, at 60 mcg/kg/hour for 0.5 to 1 hour, and at 90 mcg/kg/hour for 1 to 6 hours, on Day 1 of the Treatment Period.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Brexanolone IV infusion
  Other Names: Allopregnanolone; ZULRESSO®; SAGE-547

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of brexanolone in participants with tinnitus following a single 6-hour continuous intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Participant has a designated companion for the Clinic Treatment Visit who will drive them when they leave the clinic
2. Participant is in good physical health and has no clinically significant findings (excluding tinnitus), as determined by the investigator on medical history and physical examination, including neurologic and mental status examinations, 12-lead electrocardiogram (ECG), or clinical laboratory tests
3. Participant has a diagnosis of subjective, idiopathic, unilateral or bilateral, non-pulsatile tinnitus (e.g., not due to medical disease) of ≥6 months and <10 years duration
4. Participant has mild to severe tinnitus distress according to Tinnitus Handicap Inventory (THI) score of 24 to 68 at Screening
5. Participant is willing and able to safely discontinue the use of central nervous system (CNS) depressants (e.g., opioids and benzodiazepines), antidepressants, anticonvulsants, CNS stimulants (with the exception of caffeine), aspirin, other nonsteroidal anti inflammatory drugs, and aminoglycosides at least 14 days or 5 half-lives (whichever is longer) prior to receiving IP and through completion of the study

Exclusion Criteria:

1. Participant has history or presence of any neurologic disease or condition, including, but not limited to, unexplained loss of consciousness, seizure disorder including a prior nonfebrile seizure, and closed head trauma with clinically significant sequelae
2. Participant has a history of sleep apnea or any clinically significant respiratory conditions that may predispose the participant to hypoxia during the infusion
3. Participant intends to start or discontinue a pharmacological or nonpharmacological therapy (e.g., psychotherapy, sound therapy, masking, transcranial magnetic stimulation [TMS]) for tinnitus during the course of the study
4. Participant has currently active and medically significant or uncontrolled hepatic, renal, cardiovascular, pulmonary, gastrointestinal, hematological, immunologic, metabolic disease (hypothyroidism with stable thyroid replacement is acceptable)
5. Participant's tinnitus can be modulated by maneuvers of the temporomandibular joint, head and neck, eyes, or limbs, or otherwise attributed to somatosensory cause or has had prior otoscopic surgeries or cholesteatoma
6. Participants has current unilateral or bilateral hearing loss of 30 decibel (dB) or greater (mild hearing loss) in one or more tested frequencies (500 Hertz [Hz], 1000 Hz, 2000 Hz, and 4000 Hz), 60 dB or greater at 6000 Hz and 8000 Hz, asymmetry of 30 dB or greater in two or more tested frequencies, or uses a cochlear implant or hearing aid
7. Participant has history of chronic otitis media (>3 per year during past 5 years)
8. Participant has a total score of 15 or greater (i.e., moderately severe) on the Patient Health Questionnaire-9 (PHQ-9) at Screening
9. Participant has diagnosis of moderate or severe substance use disorder (excluding nicotine dependence) within 12 months of Screening, has a positive screen for drugs of abuse including tetrahydrocannabinol (THC) on Day 1 prior to dosing, or has a positive screen for alcohol on Day 1 prior to dosing
10. Participant has a known allergy to progesterone, allopregnanolone, or any IP excipient
11. Participant has had exposure to another investigational drug or device within 30 days or 5 half-lives of the investigational drug, whichever is longer, prior to the Day 1 visit
12. Participant has a history of suicidal behavior within 2 years or answers "YES" to Questions 3, 4, or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) at Screening or at Day 1 or is currently at risk of suicide in the opinion of the investigator
13. Participant has donated 1 or more units (1 unit = 450 milliliter [mL]) of blood or experienced acute loss of an equivalent amount of blood within 60 days prior to Day 1
14. Participant has any condition, comorbidity, or lifestyle consideration that in the opinion of the investigator would limit or interfere with the participant's ability to complete or partake in the study
15. Participant is unwilling or unable to comply with study procedures and the required training during the Baseline Period. The participant must complete 10 VAS assessments remotely prior to Day 1
16. Participant is unable to complete participation in the study, e.g., due to preplanned event including elective surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2023-11-21 (Actual); Study Completion 2023-11-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

REFERENCES:
- [Derived] Watson LS, O'Donnell P, Bankole K, Toubouti Y, Tyler RS, Johannesen JK. An open-label, proof-of-mechanism trial evaluating a neuroactive steroid GABA modulator in tinnitus. Front Neurol. 2025 Nov 18;16:1662226. doi: 10.3389/fneur.2025.1662226. eCollection 2025. PMID 41341514

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at one active clinical site in the United States from 10 May 2023 to 21 November 2023.
Pre-assignment Details: A total of 29 participants were screened, of which 10 were enrolled and treated.
Groups:
- Brexanolone: Participants received a 6-hour single continuous intravenous (IV) infusion of brexanolone at 30 micrograms per kilogram per hour (mcg/kg/hour) for 0 to 0.5 hours, at 60 mcg/kg/hour for 0.5 to 1 hour, and at 90 mcg/kg/hour for 1 to 6 hours, on Day 1 of the Treatment Period.
Period: Overall Study
Arm/Group | Brexanolone
Started | 10
Completed | 9
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety set included all participants who received any amount of brexanolone.
Groups:
- Brexanolone: Participants received a 6-hour single continuous IV infusion of brexanolone at 30 mcg/kg/hour for 0 to 0.5 hours, at 60 mcg/kg/hour for 0.5 to 1 hour, and at 90 mcg/kg/hour for 1 to 6 hours, on Day 1 of the Treatment Period.
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (9.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease temporally associated with the use of a medicinal (investigational) product whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE with onset after the start of brexanolone, or any worsening of a pre-existing medical condition/adverse event with onset after the start of brexanolone and throughout the study.
Time Frame: Up to Day 15
Population: Safety set included all participants who received any amount of brexanolone.
Measure: Count of Participants; unit: Participants
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
Participants | 1

2. Secondary Outcome: Change From Baseline (Observed Value) to Hour 6 of Infusion in Visual Analog Scale-Loudness (VAS-L) Ratings
Description: VAS-L is a subject-rated scale used to assess the perceived loudness of tinnitus. Participants answered the question "How loud is your tinnitus now?" on a horizontal scale anchored on left by "not audible" (score of 0) and on right by "extremely loud" (score of 100). Higher scores represent greater severity. Negative change from baseline represents better outcome of the treatment.
  For the treatment period (Day 1), baseline was defined as the most recent value immediately prior to the start of brexanolone infusion, or predose.
Time Frame: Baseline; 0.5, 1, 2, 3, 4, 5, and 6 hours during brexanolone infusion on Day 1
Population: Efficacy set included all participants who received any amount of brexanolone and had at least one post-baseline efficacy evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 1, Hour 0.5 | -3.1 (8.33)
  Change at Day 1, Hour 1 | -8.1 (14.13)
  Change at Day 1, Hour 2 | -7.2 (14.41)
  Change at Day 1, Hour 3 | -11.2 (14.54)
  Change at Day 1, Hour 4 | -15.4 (16.26)
  Change at Day 1, Hour 5 | -15.7 (15.72)
  Change at Day 1, Hour 6 | -12.8 (9.32)

3. Secondary Outcome: Change From Baseline (Model Based) to Hour 6 of Infusion in VAS-L Ratings
Description: VAS-L is a subject-rated scale used to assess the perceived loudness of tinnitus. Participants answered the question "How loud is your tinnitus now?" on a horizontal scale anchored on left by "not audible" (score of 0) and on right by "extremely loud" (score of 100). Higher scores represent greater severity. Negative change from baseline represents better outcome of the treatment.
  A Mixed Model Repeated Measures (MMRM) with fixed effects for baseline VAS component value and change from baseline scores as the dependent variable is used.
  For the treatment period (Day 1), baseline was defined as the most recent value immediately prior to the start of brexanolone infusion, or predose.
Time Frame: Baseline; 0.5, 1, 2, 3, 4, 5, and 6 hours during brexanolone infusion on Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 1, Hour 0.5 | -3.10 (2.486)
  Change at Day 1, Hour 1 | -8.10 (4.441)
  Change at Day 1, Hour 2 | -7.20 (4.472)
  Change at Day 1, Hour 3 | -11.20 (4.474)
  Change at Day 1, Hour 4 | -15.40 (5.043)
  Change at Day 1, Hour 5 | -15.70 (4.826)
  Change at Day 1, Hour 6 | -12.80 (3.013)

4. Secondary Outcome: Change From Baseline (Observed Value) to Hour 6 of Infusion in Visual Analog Scale-Annoyance (VAS-A) Ratings
Description: VAS-A is a subject-rated scale used to assess the tinnitus. Participants answered the question "How much is your tinnitus annoying you now?" on a horizontal scale anchored on the left by "not annoying" (score of 0) and on the right by "extremely annoying" (score of 100). Higher scores represent greater severity. Negative change from baseline represents better outcome of the treatment.
  For the treatment period (Day 1), baseline was defined as the most recent value immediately prior to the start of brexanolone infusion, or predose.
Time Frame: Baseline; 0.5, 1, 2, 3, 4, 5, and 6 hours during brexanolone infusion on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 1, Hour 0.5 | -7.6 (13.45)
  Change at Day 1, Hour 1 | -9.8 (18.74)
  Change at Day 1, Hour 2 | -16.6 (28.68)
  Change at Day 1, Hour 3 | -16.9 (20.00)
  Change at Day 1, Hour 4 | -21.3 (28.07)
  Change at Day 1, Hour 5 | -22.0 (27.71)
  Change at Day 1, Hour 6 | -22.3 (20.92)

5. Secondary Outcome: Change From Baseline (Model Based) to Hour 6 of Infusion in VAS-A Ratings
Description: VAS-A is a subject-rated scale used to assess the tinnitus. Participants answered the question "How much is your tinnitus annoying you now?" on a horizontal scale anchored on the left by "not annoying" (score of 0) and on the right by "extremely annoying" (score of 100). Higher scores represent greater severity. Negative change from baseline represents better outcome of the treatment.
  A MMRM with fixed effects for baseline VAS component value and change from baseline scores as the dependent variable is used.
  For the treatment period (Day 1), baseline was defined as the most recent value immediately prior to the start of brexanolone infusion, or predose.
Time Frame: Baseline; 0.5, 1, 2, 3, 4, 5, and 6 hours during brexanolone infusion on Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 1, Hour 0.5 | -7.60 (4.088)
  Change at Day 1, Hour 1 | -9.80 (5.193)
  Change at Day 1, Hour 2 | -16.60 (8.108)
  Change at Day 1, Hour 3 | -16.90 (5.790)
  Change at Day 1, Hour 4 | -21.30 (7.980)
  Change at Day 1, Hour 5 | -22.00 (7.882)
  Change at Day 1, Hour 6 | -22.30 (5.167)

6. Secondary Outcome: Change From Baseline (Observed Value) to Post-infusion in VAS-L Ratings Measured Via Daily Diary Over Multiple Days
Description: VAS-L is subject-rated scale used to assess perceived loudness of tinnitus. Participants answered question "How loud is your tinnitus now?" on horizontal scale anchored on left by "not audible" (score of 0) and on right by "extremely loud" (score of 100) via daily diary over multiple days. Higher scores= greater severity. Negative change from baseline= better outcome of treatment. For remote assessments (Day 2 through 7), ratings were obtained twice daily (morning and evening). Daily arithmetic mean was calculated by averaging morning and evening scores. If a participant was missing either a morning or evening score, then single available score was used as the mean for that day.
  Baseline is defined as the average value of Day -7 to Day -1 measurements. This was calculated by summing daily arithmetic means and dividing by total number of non-missing days.
Time Frame: Baseline; Days 2, 3, 4, 5, 6, and 7 after brexanolone infusion given on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 2 | -17.56 (19.125)
  Change at Day 3 | -17.51 (22.231)
  Change at Day 4 | -15.61 (20.084)
  Change at Day 5 | -16.76 (22.388)
  Change at Day 6 | -16.96 (22.235)
  Change at Day 7 | -11.31 (19.509)

7. Secondary Outcome: Change From Baseline (Model Based) to Post-infusion in VAS-L Ratings Measured Via Daily Diary Over Multiple Days
Description: VAS-L is subject-rated scale used to assess perceived loudness of tinnitus. Participants answered question "How loud is your tinnitus now?" on horizontal scale anchored on left by "not audible" (score of 0) and on right by "extremely loud" (score of 100) via daily diary over multiple days. Higher scores= greater severity. Negative change from baseline= better outcome of treatment. For remote assessments (Day 2 through 7), ratings were obtained twice daily (morning and evening). Daily arithmetic mean was calculated by averaging morning and evening scores. If a participant was missing either a morning or evening score, then single available score was used as the mean for that day. A MMRM with fixed effects for baseline VAS component value and change from baseline scores as the dependent variable is used.
  Baseline is defined as the average value of Day -7 to Day -1 measurements. This was calculated by summing daily arithmetic means and dividing by total number of non-missing days.
Time Frame: Baseline; Days 2, 3, 4, 5, 6, and 7 after brexanolone infusion given on Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 2 | -17.56 (6.769)
  Change at Day 3 | -17.51 (8.035)
  Change at Day 4 | -15.61 (6.805)
  Change at Day 5 | -16.76 (8.064)
  Change at Day 6 | -16.96 (7.721)
  Change at Day 7 | -11.31 (7.330)

8. Secondary Outcome: Change From Baseline (Observed Value) to Post-infusion in VAS-A Ratings Measured Via Daily Diary Over Multiple Days
Description: VAS-A is subject-rated scale used to assess the tinnitus. Participants answered the question "How much is your tinnitus annoying you now?" on horizontal scale anchored on left by "not annoying" (score of 0) and on right by "extremely annoying" (score of 100) via daily diary over multiple days. Higher scores=greater severity. Negative change from baseline=better outcome of treatment. For remote assessments (Day 2 through 7), ratings were obtained twice daily (morning and evening). Daily arithmetic mean was calculated by averaging morning and evening scores. If a participant was missing either a morning or evening score, then single available score was used as the mean for that day.
  Baseline is defined as the average value of Day -7 to Day -1 measurements. This was calculated by summing daily arithmetic means and dividing by total number of non-missing days.
Time Frame: Baseline; Days 2, 3, 4, 5, 6, and 7 after brexanolone infusion given on Day 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 2 | -19.41 (19.492)
  Change at Day 3 | -16.01 (21.161)
  Change at Day 4 | -13.41 (23.037)
  Change at Day 5 | -15.16 (26.075)
  Change at Day 6 | -11.51 (27.493)
  Change at Day 7 | -7.61 (23.659)

9. Secondary Outcome: Change From Baseline (Model Based) to Post-infusion in VAS-A Ratings Measured Via Daily Diary Over Multiple Days
Description: VAS-A is subject-rated scale used to assess the tinnitus. Participants answered the question "How much is your tinnitus annoying you now?" on horizontal scale anchored on left by "not annoying" (score of 0) and on right by "extremely annoying" (score of 100) via daily diary over multiple days. Higher scores=greater severity. Negative change from baseline=better outcome of treatment. For remote assessments (Day 2 through 7), ratings were obtained twice daily (morning and evening). Daily arithmetic mean was calculated by averaging morning and evening scores. If a participant was missing either a morning or evening score, then single available score was used as the mean for that day. A MMRM with fixed effects for baseline VAS component value and change from baseline scores as the dependent variable is used.
  Baseline is defined as the average value of Day -7 to Day -1 measurements. This was calculated by summing daily arithmetic means and dividing by total number of non-missing days.
Time Frame: Baseline; Days 2, 3, 4, 5, 6, and 7 after brexanolone infusion given on Day 1
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Brexanolone
Number analyzed (Participants) | 10
score on a scale
  Change at Day 2 | -19.41 (7.266)
  Change at Day 3 | -16.01 (8.111)
  Change at Day 4 | -13.41 (8.288)
  Change at Day 5 | -15.16 (8.716)
  Change at Day 6 | -11.51 (9.523)
  Change at Day 7 | -7.61 (8.078)

ADVERSE EVENTS:
Time Frame: Up to Day 15
Description: Safety set included all participants who received any amount of brexanolone.
Arm/Group | Brexanolone
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brexanolone (N=10)
Tinnitus (Ear and labyrinth disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT05645432/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT05645432/SAP_001.pdf